CLINICAL TRIAL: NCT01545973
Title: Measuring Skin Electrical Potential With the Kelvin Probe: Underlying Physiology
Brief Title: Understanding the Physiological Implications of Scanning Kelvin Probe Measurements
Status: Suspended | Type: Observational
Why Stopped: Repair of minor software glitches
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew A. Ahn, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 55R21AT005249-02
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Individuals; Skin Electrical Potential

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Human subjects without chronic medical conditions, defined as conditions requiring chronic medication use.
  Interventions: Other: Skin Moistening, Skin Denuding

INTERVENTIONS:
Other: Skin Moistening, Skin Denuding — Application of normal saline to skin and Tape stripping of the superficial skin

SUMMARY:
The purpose of this study is to evaluate the effects of skin thickness, skin moisture, and sweat gland density on Scanning Kelvin Probe measurements.

DETAILED DESCRIPTION:
The Scanning Kelvin Probe measures the electrical potential of material surfaces without actually touching it. Although this technology has been applied to non-living materials (e.g. metal and semiconductors) before, it has not been effectively applied to biological materials, much less to live human skin . This project aims to evaluate the use of Scanning Kelvin Probe to live human skin by investigating the effects of skin thickness, skin moisture, and sweat glands on Kelvin Probe measurements of electrical potential. Testing will be performed on the arms and hands of twenty four healthy individuals under different study conditions.

ELIGIBILITY:
Inclusion Criteria:

* "Healthy" is defined as not having a chronic medical condition requiring daily medications (hypertension, diabetes, hypothyroidism, etc)

Exclusion Criteria:

* autonomic disorders (sweating irregularities), skin disorders, extensive burns/scars on the hand, tremors, neuromuscular conditions, restless leg syndrome, movement disorders, and implanted cardiac defibrillator/pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Surface Electrical Potential | 1 day
  The electrical potential of skin obtained from the Scanning Kelvin Probe

SECONDARY OUTCOMES:
Electrical Impedance | One day
  Electrical impedance (measurement) obtained through another, more conventional measurement device.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C. Ahn, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States